CLINICAL TRIAL: NCT00119730
Title: Abbreviated Fludarabine / Mitoxantrone / Rituximab Chemotherapy Followed by Zevalin for Relapsed Mantle Cell Lymphoma
Brief Title: Chemotherapy Followed by Zevalin for Relapsed Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Biogen (Industry)
Responsible Party: Principal Investigator, Jennifer R. Brown, MD, PhD, Assistant Professor of Medicine, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-251
Record Dates: First submitted 2005-07-07; First posted 2005-07-14 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Mantle Cell Lymphoma
Keywords: Fludarabine; Mitoxantrone; Rituximab; Zevalin; Mantle Cell Lymphoma; Relapsed Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — fludarabine; fludarabine phosphate; Mitoxantrone; Rituximab; ibritumomab tiuxetan

ARMS (1):
- Fludarabine, Mitoxantrone, Rituximab, Zevalin (Experimental): Drug: Fludarabine Given on days 1-3 of each 28-day cycle Drug: Mitoxantrone Given on day 1 of each 28-day cycle Drug: Rituximab Given on day 1 of each 28-day cycle Drug: Zevalin Given after two cycles if there is no disease progression.
  Interventions: Drug: Fludarabine; Drug: Mitoxantrone; Drug: Rituximab; Drug: Zevalin

INTERVENTIONS:
Drug: Fludarabine — Given on days 1-3 of each 28-day cycle
  Other Names: Fludara
Drug: Mitoxantrone — Given on day 1 of each 28-day cycle
  Other Names: Mitozantrone
Drug: Rituximab — Given on day 1 of each 28-day cycle
  Other Names: Rituxan, MabThera and Zytux
Drug: Zevalin — After two cycles if there is no disease progression, zevalin treatment will be given. Rituximab will be given followed by an imaging dose of zevalin. Two or three scans will be performed over a week to determine if it is safe to give the full treatment dose of zevalin. The treatment dose is given with the second infusion or rituximab, seven days after the first dose.
  Other Names: Ibritumomab tiuxetan

SUMMARY:
* The purpose of this study is to find out whether combining a short course of chemotherapy (Fludarabine, Mitoxantrone and Rituximab) followed by Zevalin will be effective in treating relapsed mantle cell lymphoma.
* The secondary purposes of the study are to determine the safety and to evaluate whether there is additional benefit from Zevalin therapy following the chemotherapy.

DETAILED DESCRIPTION:
* Patients receive fludarabine (days 1-3), mitoxantrone (day 1), and rituximab (day 1) of each 28-day cycle.
* Patients undergo a CT scan and bone marrow biopsy after two cycles. Unless the cancer has progressed, the patient will then receive Zevalin study treatment.
* Blood counts are taken every week for 12 weeks. After 12 weeks, a CT scan and bone marrow biopsy are performed.
* Long-term followup is 4 years. Physical exam and blood work is performed every 3 months for the first two years. Following that, physical exams and blood work is every 6 months for another two years. CT scans and bone marrow biopsies are every 6 months during this 4 year followup period.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed mantle cell lymphoma in 1st or 2nd relapse, or with persistent disease following induction therapy.
* Measurable disease (lymph node > 1.5 cm)
* No anti-cancer therapy for three weeks (six weeks if Rituximab, nitrosourea or Mitomycin C) prior to study initiation, and fully recovered from all toxicities associated with prior surgery, radiation treatments, chemotherapy, or immunotherapy
* An IRB-approved signed informed consent
* Age >/= 18 years
* Expected survival >/= 3 months
* ECOG performance status 0, 1, or 2
* Acceptable hematologic status within two weeks prior to registration, including: * Absolute neutrophil count ([segmented neutrophils + bands] x total WBC) ≥ 1,500/mm3; * Platelet counts ≥ 100,000/mm3
* Female patients who are not pregnant or lactating
* Men and women of reproductive potential who are following accepted birth control methods (as determined by the treating physician, however abstinence is not an acceptable method)
* Patients previously on Phase II drugs if no long-term toxicity is expected, and the patient has been off the drug for eight or more weeks with no significant post treatment toxicities observed

Inclusion Criteria for Proceeding with Zevalin:

* Hematologic recovery from FMR (ANC >1500, platelets > 100,000)
* Stable or responding disease on restaging following two cycles of FMR
* < 25% of bone marrow cellularity involved with lymphoma on restaging bone marrow biopsy
* Bone marrow cellularity at least 20% (including lymphoma and normal cells)
* Total bilirubin < 2.0 mg/dL (if total bilirubin is >75% indirect, then may use direct bilirubin < 0.8 mg/dL)
* Serum creatinine < 2.0 mg/dL
* No G-CSF or GM-CSF therapy within two weeks prior to Zevalin treatment, or neulasta within four weeks prior to Zevalin treatment
* No evidence of altered biodistribution of 111-In-Zevalin as indicated by:

  1. Absent cardiac blood pool on day 1, with high liver / spleen uptake
  2. Lung uptake greater than blood pool on day 1 or greater than liver on day 2-3
  3. Kidney (in posterior view) or bowel uptake greater than liver on day 2-3

Exclusion Criteria:

* Patients with impaired bone marrow reserve, as indicated by one or more of the following: * Prior myeloablative therapies with allogeneic or autologous bone marrow transplantation (ABMT) or peripheral blood stem cell (PBSC) rescue; * Platelet count < 100,000 cells/mm3; * Prior external beam radiation to >25% of active bone marrow; * History of failed stem cell collection
* Prior radioimmunotherapy
* Known cardiac ejection fraction < 40%. In patients with prior adriamycin exposure >= 300 mg/m2, echocardiogram must be obtained within three months prior to registration
* Known CNS lymphoma (lumbar puncture only required if symptomatic)
* Chronic lymphocytic leukemia (CLL)
* HIV or AIDS-related lymphoma
* Pleural effusion or ascites
* Abnormal liver function: total bilirubin > 2.0 mg/dL (if total bilirubin is >75% indirect, then may use direct bilirubin > 0.8 mg/dL)
* Abnormal renal function: serum creatinine > 2.0 mg/dL
* G-CSF or GM-CSF therapy within two weeks prior to treatment, or neulasta within four weeks
* Positive direct antiglobulin test
* Major surgery, other than diagnostic surgery, within four weeks
* Serious nonmalignant disease or infection which in the opinion of the investigator would compromise protocol objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-02; Primary Completion 2006-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine the response rate to two cycles of FMR + Zevalin in patients with relapsed mantle cell lymphoma, using a two-stage design. | 2 years

SECONDARY OUTCOMES:
To describe the progression-free survival
To determine the safety of FMR + Zevalin in these subjects | 2 years
To determine the impact of Zevalin on minimal residual disease in subjects with relapsed mantle cell lymphoma | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R Brown, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts